CLINICAL TRIAL: NCT06334185
Title: Evaluation of Vaccination for Streptococcus Pneumoniae in Adults With an Episode of Invasive Pneumococcal Infection: a Retrospective Study in Two Lombardy Centers in the Pre-pandemic Phase From 2015 to 2019.
Brief Title: Evaluation of Vaccination for Streptococcus Pneumoniae in Adults With an Episode of Invasive Pneumococcal Infection.
Acronym: pVax
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Lecco (Other)
Collaborators: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Stefania Piconi, Director of Infectious Diseases Unit, Azienda Ospedaliera di Lecco
Other Study IDs: pVax
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Invasive Pneumococcal Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Respiratory tract infections are among the leading causes of death worldwide and many of these infections are preventable through vaccination. One of the most important bacteria from an etiological and mortality point of view regarding respiratory and systemic infections is the gram-positive Streptococcus pneumoniae. Four types of vaccines are currently available for this pathogen: three pneumococcal conjugate vaccines (PCV13, PCV15, and PCV20) and one polysaccharide vaccine (PPSV23). In Italy, people over 65 years of age and people suffering from chronic pathologies with effects on the immune system would be advised to be vaccinated with the pneumococcal conjugate vaccine and with the polysaccharide vaccine as a second dose.

However, there are no data available in Italy on vaccination coverage in these population categories and above all the vaccination rates in patients who have a history of an episode of invasive pneumococcal infection are not known. The aim of the study is to measure how many patients are vaccinated for S. pneumoniae after hospitalization for a systemic pneumococcal infection in order to understand patients' awareness of preventing this infection after receiving a first diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old;
* Patients hospitalized at the Manzoni Hospital in Lecco or at the San Raffaele Hospital in Milan with invasive pneumococcal infection in the period between 01/01/2015 and 31/12/2019;
* Presence of a positive culture test for S. pneumoniae on blood cultures and/or liquor;
* Patients whose discharge letter or clinical documentation relating to the infectious episode is available;
* Patients whose vaccination record can be consulted (on paper or on SIAVR) and whose vaccination history is available before and after hospitalization.

Exclusion Criteria:

* Patients with positive urinary antigen for S. pneumoniae as the only microbiological finding;
* Patients whose vaccination history or vaccination records are not available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A retrospective multicenter study is planned on patients admitted to the Alessandro Manzoni Hospital in Lecco and the San Raffaele Hospital in Milan with a diagnosis of systemic pneumococcal infection from 01/01/2015 to 12/31/2019 before the SARS pandemic -CoV-2.
  All patients admitted with a diagnosis of invasive pneumococcal infection defined by positive blood or CSF cultures for S. pneumoniae by the microbiology laboratory were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of antipneumococcal vaccination in hospitalized patients for invasive pneumococcal infection between 2015 and 2019. | The information regarding vaccination after the infectious episode will be assessed by consulting the SIAVR portal or the vaccination booklet in a period between at least one month from discharge and up to 06/30/2023.

SECONDARY OUTCOMES:
Rate of pneumococcal serotype that caused the invasive infection in patients vaccinated prior to the infectious event | The information regarding vaccination after the infectious episode will be assessed by consulting the SIAVR portal or the vaccination booklet in a period between at least one month from discharge and up to 06/30/2023.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Castagna, Prof, Principal Investigator — IRCCS Ospedale San Raffaele Turro - Milano Infectious Diseases Unit